CLINICAL TRIAL: NCT00286065
Title: Multi-Centre Placebo-Controlled Randomized 2 Part Study to Determine Efficacy and Safety of Inhaled AeroLEF in the Treatment of Acute Post-Op Pain in Adult Patients Undergoing Elective Orthopedic Surgery
Brief Title: Study to Determine Efficacy and Safety of Inhaled AeroLEF in the Treatment of Acute Post-op Pain in Adult Patients Undergoing Elective Orthopedic Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: YM BioSciences (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DLXLEF-AP4
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Pain
Keywords: Pain; Fentanyl; Analgesics; Opioid; Inhalation
MeSH Terms: conditions — Pain; Respiratory Aspiration

INTERVENTIONS:
Drug: AeroLEF

SUMMARY:
The purpose of this study is to determine the effect of pain relief with AeroLEF in adult patients, following orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* male and female 18 to 70 years
* patient alert and capable of self-administering an opioid anaglesic
* Patient is scheduled for orthopedic surgery under general anesthesia
* Patient has normal laboratory values
* Physical examination with no clincially relevant findings
* Patient in general good health based on medical history and clincially acceptable
* Patient is able to understand the requirements of the study
* Patient is able to communicate effectively with study personnel _Patient voluntarily gives written approval.

Exclusion Criteria:

* During Part 2 (randomized period) which involves the use of placebo, patients who are undergoing a major orthopedic procedure that normally requires multimodal analgesia to achieve adequate postoperative pain control (e.g. major spine surgery, total knee arthoplasty) will be excluded.
* Patient is taking opioid or non-opioid analgesics on a chronic basis at doses which in the opinion of the investigator would interfere with evaluations of post-operative fentanyl efficacy.
* History of pulmonary, cardiovascular, neurologic, endocrine, hepatic, gastrointestinal (GI), or kidney disease or therapy that would jeopardize the patient's well-being by participation in this study.
* Patient has documented or self-reported medical history of sleep apnea.
* Patient has a documented hypersensitivity to fentanyl or other opioid analgesics.
* Patient has a documented hypersensitivity/allergy to the components of the liposomes used in the AeroLEF formulation, including hypersensitivity to soya lecithin or related food products such as soya bean and peanut.
* Patient is currently receiving treatment, or has received treatment in the previous two weeks, with monoamine oxidase inhibitors.
* Patient has a history of malignancy within the past 5 years, with the exception of successfully treated non?metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix.
* Patient was dosed with another investigational drug within 30 days prior to the Screening Visit.
* Patient has current therapy with CNS-depressant medications (other than stable doses of analgesics and drugs used with surgical anesthesia).
* Patient has current evidence of alcohol abuse (regularly drinks more than 4 units of alcohol per day; 1 unit = ½ pint of beer, 1 glass of wine, or 1 ounce of spirit).
* Patient has a history of abuse of licit or illicit drug substances.
* Patient, who in the opinion of the Investigator, is mentally or emotionally unsuitable to participate, or unable/unwilling to comply with the study assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123
Dates: Start 2006-01

PRIMARY OUTCOMES:
- Summed Pain Relief plus Pain Intensity Difference (SPRID) scores during the interval from Baseline post-surgery to 4 hours after the initial dose following surgery

SECONDARY OUTCOMES:
Sum of the Pain Intensity Difference scores (SPID) for 4 hours after the start of the initial dose
Sum of the Pain Relief scores (TOTPAR) for the 4 hours following the start of the initial dose
Total use of rescue analgesic drug.
Time to effective pain relief (measured by stopwatch).
Duration of effective pain relief as measured by the interval between time to onset of effective pain relief and time to first use of rescue drug (both measured by stopwatch) or next dose of study drug.
Clinician Global Impression (CGI) scores at 4 and 12 hours after the start of the initial post-surgery dose of study drug.
Patient Treatment Satisfaction Rating scores at 4 and 12 hours after the start of the initial post-surgery dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, M.D., Principal Investigator — University Health Network, Toronto; Kenneth Chisholm, M.D, Principal Investigator — Queen Elizabeth II Infirmary
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada